CLINICAL TRIAL: NCT05344183
Title: Immediate and Short-term Effects of Low-level Laser on the Functional Performance of the Lower Limbs of Jumping Athletes
Brief Title: Immediate and Short-term Effects of Low-level Laser
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Amapá (Other)
Responsible Party: Principal Investigator, Renan Lima Monteiro, Clinical Professor, Universidade Federal do Amapá
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 120422
Record Dates: First submitted 2022-04-12; First posted 2022-04-25 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Fatigue; Muscle Injury
MeSH Terms: conditions — Fatigue | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lasertherapy (Experimental)
  Interventions: Device: Low-level laser
- Sham lasertherapy (Sham Comparator)
  Interventions: Device: Low-level laser

INTERVENTIONS:
Device: Low-level laser — A laser will be used in the quadriceps and gluteus medius muscles with the following parameters described for muscle recovery: dose of 40 J for the gluteus medius muscle, 180 J for the quadriceps muscle; power from 50 to 200 mW per diode (for single probes), 10 to 35 mW per diode (for cluster probes). The full power of the device cannot lead to thermal effects; Wavelengths of 950 nm (infrared).

SUMMARY:
Athletes experience an exhaustive routine of training, associated with the reduced time of rest, facilitates the appearance of muscle fatigue, which increases the risk of muscle injuries, especially during the execution of the jump. Low Level Lasertherapy is a technique that has been increasingly improved due to the physiological effects it provides in the muscle recovery process. However, there is still a lack of studies focused on the use of this technique in functional improvement, especially in jumping sports. Objectives: To evaluate the immediate and short-term effects of low-level laser on the functional performance of lower limbs of jumping athletes and to evaluate the short-term effects of low-level laser on the activation of the gluteus medius and quadriceps muscles. Methods: This is a brief, double-blind, randomized, placebo-controlled clinical trial. Will be recruited 24 handball and volleyball players aged between 18 to 35 years. The primary outcome of our study is functional performance (modified hop test and modified SEBT), and as a secondary outcome (level of electromyographic activity). After the baseline assessments, the athletes will be randomized and allocated into two groups: Intervention Group (IG, n=12) and Control Group (CG, n=12) and submitted to a fatigue protocol, followed by laser therapy or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Handball and volleyball athletes;
* Age between 18 and 35 years;
* Both sexes;
* Athletes who maintain a training routine for their sport, at least twice a week

Exclusion Criteria:

* History of acute injury to the lower limbs (LL) in the last 2 months;
* Occurrence of pain and injury during the study;
* Any change in physical activity routine during the week of assessments.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-09-03 (Actual); Primary Completion 2023-11-12 (Actual); Study Completion 2024-12-12 (Estimated)

PRIMARY OUTCOMES:
Functional Performance | 6 days
  For the evaluation of the functional performance, the tests will be used is the horizontal unipedal jump.

SECONDARY OUTCOMES:
Muscle activity | 2 days
  Muscle activations will be collected using a FREEEMG 1000 electromyographic instrument in the quadriceps femoris muscles.

CONTACTS AND LOCATIONS:
Locations (1):
- Renan Lima Monteiro, Macapá, Amapá, Brazil

IPD SHARING:
Plan to Share IPD: Undecided